CLINICAL TRIAL: NCT03381079
Title: Posterior Scleral Reinforcement for Adults With High Myopia
Brief Title: Efficacy and Safety of Posterior Scleral Reinforcement on Controlling Myopia in Adults With High Myopia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Shi-Ming Li, Vice director of Ophthalmology clinical research center, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRECKY2017-049
Record Dates: First submitted 2017-12-12; First posted 2017-12-21 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: High Myopia; Posterior Scleral Reinforcement; Adults; Axial Elongation; Myopia Progression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical group (Experimental): In this arm, the adults with high myopia will be given posterior scleral reinforcement.
  Interventions: Procedure: Posterior scleral reinforcement
- Control group (No Intervention): In this arm, the adults with high myopia will not be given any surgical treatment.

INTERVENTIONS:
Procedure: Posterior scleral reinforcement — Posterior scleral reinforcement (pPSR) is a procedure applied with autologous or biological material or synthetic materials reinforcing pole of the sclera after eyeball, in order to prevent or alleviate myopic development.
  Arms: Surgical group

SUMMARY:
This study will evaluate the efficacy and safety of posterior scleral reinforcement on controlling myopia progression, including change in refraction, axial elongation as well as sight-threatening complications, in adults with high myopia. Half the adults will receive posterior scleral reinforcement, while the other half will receive no surgerical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cycloplegic spherical equivalent less than -6.0 D
* Myopia progression greater than 1.0 D per year
* Normal IOP, no strabismus or any other ocular pathological changes
* no any other ocular or systematic diseases that may affect refractive development

Exclusion Criteria:

* Currently or history using other interventions to control myopia progression (acupuncture, drugs, contact lens, ear needles and so on)
* Unable to cooperate with the ocular examination,questionnaire survey,or orthokeratology wearing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic autorefraction | 2 years
  Level of myopia and myopia progression as assessed by autorefraction
Axial length | 2 years
  Longth of the eyeball as assessed by IOL Master or Lenstar

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 2 years
  Bleeding, inflammation or retinal detachment as assessed by B scan, slitlamp, etc.
Visual acuity | 2 years
  An index for visual function measured by visual acuity chart

CONTACTS AND LOCATIONS:
Overall Officials: Ningli Wang, PhD, Study Chair — Beijing Tongren Eye Center, Beijing Tongren Hospital

IPD SHARING:
Plan to Share IPD: Undecided